CLINICAL TRIAL: NCT00223730
Title: Chemotherapy Toxicity Reduction Via Urea Cycle Support
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Brian Christman, Professor of Medicine and Principal Investigator, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 990675; NIH HL-55198 (Other: NIH); NIH 1P-30CA68485 (Other: NIH); NIH 1RO1-CA092313-01 (Other: NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cancer
Keywords: Peripheral Blood Stem Cell Transplant; Bone Marrow Transplant; Citrulline; Urea Cycle; Hepatic Injury; Allogeneic PBSCT; Matched-Unrelated PBSCT
MeSH Terms: conditions — Neoplasms | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- citrulline (Experimental): Patients randomized to receive oral citrulline at 3.8 gm/m2 in split BID dosing
  Interventions: Drug: Citrulline
- Placebo (Placebo Comparator): Patients randomized to receive oral diluent for citrulline in BID dosing
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citrulline — Oral provision of amino acid citrulline to support impaired urea cycle function during escalated dose chemotherapy for stem cell transplant
  Arms: citrulline
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patients undergoing bone marrow transplantation (BMT) and peripheral blood stem cell transplants (PBSCT) frequently develop organ dysfunctions, much of which may be initiated by damage to the liver and to cells lining blood vessels.

We, the researchers at Vanderbilt University, propose to perform a randomized, prospective, double-blind, placebo-controlled study of 144 patients undergoing allogeneic marrow transplantation. The treatment is aimed at supporting hepatic urea cycle function in patients receiving escalated dose chemotherapy/BMT. By so doing we hope to prevent development of hepatic venoocclusive disease (HVOD) and acute lung injury (ALI), two morbid complications of BMT. Patients will be randomized to receive oral citrulline, a urea cycle amino acid intermediate, or placebo beginning before conditioning therapy and continuing until 21 days after BMT. All patients will be followed for 100 days after study enrollment with intensive data collection.

ELIGIBILITY:
Inclusion Criteria:

* We propose to study 144 patients undergoing allogeneic bone marrow transplantation or peripheral blood stem cell transplant over a 4 year period.
* Patients of either sex and of any race or ethnic origin, older than age greater than or equal to13, and admitted to the Myelosuppression Unit (MSU) of Vanderbilt University Hospital or the VA Hospital to undergo bone marrow transplantation will be recruited for this study.

Exclusion Criteria:

* Patients will be excluded if pregnant (unlikely) or if informed consent cannot be obtained.
* Because of the intrinsic toxicity of the treatment regimens, BMT is not usually offered to patients with severe underlying derangements in organ function. Nevertheless, other exclusions that will prevent entry of patients into the study include advanced renal or hepatic failure (serum creatinine > 6mg/dl, serum bilirubin >3.5 mg/dl), moribund patients, and patients whose primary physician is not committed to full support of the patient (i.e. "Do Not Resuscitate").
* Other exclusions will include patients enrolled in another experimental (interventional) protocol aimed at reducing transplant related complications during BMT, patients testing positive for HIV, those who have had previous BMT, and patients actively bleeding at the time of initiation of induction therapy. We will not exclude patients undergoing newer regimens of cytotoxic chemotherapy.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian W. Christman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States